CLINICAL TRIAL: NCT04404192
Title: A Phase 2a Double-blind, Placebo-controlled, Parallel Study of PH94B Nasal Spray in the Treatment of Adjustment Disorder With Anxiety
Brief Title: PH94B in the Treatment of Adjustment Disorder With Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH94B-CL029
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Adjustment Disorder With Anxious Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PH94B (Experimental): Intranasal spray 3.2 micrograms four times a day for 28 days
  Interventions: Drug: PH94B
- Placebo (Experimental): Intranasal spray four times a day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PH94B — Intranasal administration of 100 microliters to each nostril 4 times a day
  Other Names: Aloradine
  Arms: PH94B
Drug: Placebo — Intranasal administration of 100 microliters to each nostril 4 times a day.
  Arms: Placebo

SUMMARY:
This placebo-controlled clinical study is designed to evaluate the efficacy, safety and tolerability of administration of PH94B nasal spray four times per day as a treatment of Adjustment Disorder with Anxiety symptoms in adults. Subject participation in the Study will last a total of 6 to 10 weeks, depending on the duration of the screening period and whether they need a washout of concomitant anxiolytics. Upon signing an investigation review board approved informed consent, all subjects will complete Visit 1 (Screening) and enter a screening period lasting 7 to 35 days that could include taper of concomitant anxiolytics, if necessary. Screening visit will consist of safety assessments (medical history, physical examination, laboratory samples, electrocardiogram, urine drug screen, and urine pregnancy test [if appropriate]) and psychiatric assessments to determine eligibility. Subjects will then return to complete Visit 2 (Baseline). If the subject continues to meet inclusion and exclusion criteria, the subject will be randomized 1:1 to PH94B or placebo. Subjects will then commence 4 weeks of double-blind treatment with randomized investigational product (PH94B or placebo) four times per day.

Subjects will return for weekly site visits (Visits 3, 4, 5, and 6), in which the subject will return the vial dispensed at the previous visit and receive a new vial, except at Visit 6 in which no new vial will be dispensed. Changes in AEs and concomitant medications will be collected. During these visits, psychiatric scales will be completed. When the subject returns for Visit 6, besides the assessments completed at Visits 3 through 5, the subjects will complete a brief physical examination, electrocardiogram, laboratory tests (chemistry and blood), and urinalysis. Any remaining IP vials will be collected. The subject will then come back after a one week washout period for Follow-up visit (Visit 7).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided prior to conducting any study-specific assessment.
2. Male and female adults, 18 through 65 years of age, inclusive.
3. Current diagnosis of AjDA as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition.
4. Clinician-rated Hamilton Anxiety Scale (HAM-A) score ≥20 at Screening (Visit 1) and no greater than 15% decrease at Baseline (Visit 2).
5. Clinician-rated Hamilton Depression Scale (HAM-D) total score <18 at Screening (Visit 1) and Baseline (Visit 2).
6. Clinical Global Impression - Severity Scale (CGI-S) score ≥4 at both Screening (Visit 1) and Baseline (Visit 2)
7. Women of child bearing-potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the Study, and must also have a negative urine pregnancy test result at both Screening (Visit 1) and Baseline (Visit 2), prior to investigational product (IP) administration. Effective methods of contraception include: condoms with spermicide, diaphragm with spermicide, hormonal contraceptive agents (oral, transdermal, or injectable), or implantable contraceptive devices.
8. Males whose sexual partners are women of childbearing potential must commit to the consistent and correct use of an effective method of birth control throughout the study.
9. Negative COVID-19 test either in the presence of COVID-19 symptoms or after exposure to someone with a positive COVID-19 test.

Exclusion Criteria:

1. Any history of schizophrenia or schizoaffective disorder.
2. Any other current Axis I disorder, including, but not limited to, major depressive disorder, bipolar disorder, post-traumatic stress disorder, obsessive-compulsive disorder, premenstrual dysphoric disorder, and generalized anxiety disorder, which is in poor control and the primary focus of treatment.
3. A diagnosis of social anxiety disorder with a score >60 on the Liebowitz Social Anxiety Scale.
4. Subjects who meet criteria for moderate or severe alcohol or substance use disorder within the 1 year prior to Study entry.
5. In the opinion of the investigator, the subject has a significant risk for suicidal behavior during the course of their participation in the study, or considered to be an imminent danger to themselves or others.
6. Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, anosmia, or nasal septum perforation that may have damaged the nasal chemosensory epithelium.
7. An acute or chronic condition, including an infectious illness, uncontrolled seasonal allergies at the time of the study, or significant nasal congestion that potentially could affect drug delivery to the nasal chemosensory epithelium. The Investigator may allow concomitant use of over-the-counter nasal decongenstants as needed, since there is no apparent drug interaction between these and PH94B.
8. Concomitant use of any anxiolytics, such as benzodiazepines or buspirone, during the Study and within 30 days of Baseline (Visit 2).
9. Concomitant use of any over-the-counter, prescription product, or herbal preparation for treatment of the symptoms of anxiety during the Study and within 30 days before Study entry. Selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, or other approved antidepressants are permitted as long as the dose has been stable for 30 days prior to Baseline (Visit 2).
10. Women who have a positive urine or serum pregnancy test at either Screening or Baseline visit or are currently breast feeding.
11. Subjects with clinically significant abnormalities in hematology, blood chemistry, urinalysis, electrocardiogram, or physical examination identified at the Screening visit that in the clinical judgment of the Investigator, could place the subject at undue risk, interfere with study participation, or confound the results of the study.
12. Subjects with a positive urine drug screen at either the Screening visit or Baseline visit (not including tetrahydrocannabinol).
13. Any current clinically significant and/or uncontrolled medical condition, based on medical history or as evidenced in screening assessments, such as SARS-Cov-2, HIV, cancer, stroke, congestive heart failure, uncontrolled diabetes mellitus, or any other medical condition or disease that, in the clinical judgment of the Investigator, could place the subject at undue risk, interfere with Study participation, or confound the results of the Study.
14. Use of a concomitant medication that, in the clinical judgement of the Investigator, could place the subject at undue risk, interfere with study participation, or confound the results of the study.
15. History of cancer or malignant tumor not in remission for at least 2 years. Basal cell skin cancers are not exclusionary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VistaGen Clinical Site, Watertown, Massachusetts
  - VistaGen Clinical Site, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PH94B: PH94B Nasal Spray - 3.2 micrograms four times a day for 28 days
- Placebo: Placebo Nasal Spray - four times a day for 28 days
Period: Overall Study
Arm/Group | PH94B | Placebo
Started | 19 | 22
Completed | 15 | 19
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Missed 2 or more consecutive visits during 4-week treatment period | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PH94B | Placebo | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (12.74) | 41.5 (13.00) | 38.8 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 41
Hamilton Anxiety Scale (HAM-A) Total Score [Mean (Standard Deviation); unit: score on a scale] — The HAM-A questionnaire consists of 14 items, each scored on a 5-point scale (0="Not present", 1="Mild", 2="Moderate", 3="Severe", 4="Very severe. The HAM-A total score is calculated as the sum of the 14 individual scores, ranging from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe.
  score on a scale | 23.7 (3.32) | 23.1 (2.64) | 23.4 (2.95)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Scale (HAM-A) Score
Description: Least squares mean change from baseline to Visit 6 in anxiety level as measured by the HAM-A at the end of the 4-week treatment period. The HAM-A questionnaire consists of 14 items, each scored on a 5-point scale (0="Not present", 1="Mild", 2="Moderate", 3="Severe", 4="Very severe. The HAM-A total score is calculated as the sum of the 14 individual scores, ranging from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity, and 25-30 moderate to severe. Higher total scores indicate more severe disease.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 19 | 22
score on a scale | -12.5 (1.31) | -12.6 (1.22)
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = 0.9338, ANCOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-3.5 to 3.8], Standard Error of Mean 1.79

2. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement Rating (CGI-I) Response
Description: The CGI-I scale is a clinician-rated scale to assess illness improvement. The CGI-I scale includes one item scored from 1 (Very much less anxious) to 7 (Very much more anxious) with 4 being no change. Subjects are considered CGI-I responders with scores of 1 (Very much less anxious) or 2 (Much less anxious).
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 12 | 16
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = 0.3720, Wald Normal Approximation [Z]; Odds Ratio (OR) = 0.5358, 95% CI 2-sided [0.1361 to 2.1086]

3. Secondary Outcome: Percentage of Participants With Patient Global Impression of Change (PGI-C) Response
Description: The PGI-C is a self-administered instrument that measures change in subjects' overall improvement with treatment on a scale where 1= "very much improved" and 7= "very much worse". Values for comparison were the proportion of "responders" in each group, defined as subjects receiving scores of 1 (very much improved) or 2 (much improved) at the end of treatment.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 8 | 14
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = 0.1230, Wald Normal Approximation [Z]; Odds Ratio (OR) = 0.3637, 95% CI 2-sided [0.1006 to 1.3152]

4. Secondary Outcome: Adjustment Disorder New Module Scale (ADNM) Score
Description: Least squares mean change from baseline to Visit 6 in ADNM total score. THE ADNM consists of 18-item stressful life checklist and a list of 20 statements about which reactions these types of events can trigger. Subjects are asked to indicate of how often the statements apply on a 4-point scale (1= "never", 2= "rarely", 3= "sometimes", 4= "often"). ADNM total score is calculated as the sum of the 20 frequency scores. Higher total scores indicate more severe disease.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 19 | 22
score on a scale | -9.9 (2.19) | -12.1 (2.13)
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = 0.4764, ANCOVA; LS Mean Difference = 2.2, 95% CI 2-sided [-4.0 to 8.4], Standard Error of Mean 3.06

5. Secondary Outcome: International Adjustment Disorder Questionnaire (IADQ) Score
Description: Least squares mean change from baseline to Visit 6 in IADQ total score. The preoccupation, failure to adapt, and functional impairment subscale items are scored on a 5-point scale (0="Not at all", 1="A little bit", 2="Moderately", 3="Quite a bit", and 4="Extremely"). The IADQ total score is calculated as the sum of the 6 preoccupation and failure to adapt items. Higher total scores indicate more severe disease.
Time Frame: 28 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PH94B | Placebo
Number analyzed (Participants) | 19 | 22
score on a scale | -9.0 (1.49) | -11.4 (1.45)
Statistical Analysis 1: Comparison: PH94B vs Placebo; Test type: Superiority; p = 0.241, ANCOVA; LS Mean Difference = 2.5, 95% CI 2-sided [-1.7 to 6.7], Standard Error of Mean 2.08

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | PH94B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 11/19 | 11/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PH94B (N=19) | Placebo (N=22)
Headache (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1
Change in sustained attention (Psychiatric disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Oral contusion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT04404192/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT04404192/SAP_001.pdf